CLINICAL TRIAL: NCT01726920
Title: A Phase III, Multicenter, National, Open, Randomized, Parallel and Comparative Study to Evaluate the Efficacy and Safety of a Fixed-dose Combination of Naratriptan 2,5 mg + Naproxen 500 mg for the Acute Treatment of Migraine.
Brief Title: Efficacy and Safety of a Fixed-dose Combination of Naratriptan and Naproxen in Acute Treatment of Migraine.
Acronym: Copérnico
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to budget limitations, the company decided to withdraw this study.
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-NRP-03(04/12)
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Migraine; Headache
Keywords: Migraine; Naratriptan; Naproxen
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — naratriptan; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- naratriptan + naproxen (Experimental): Fixed-dose combination of naratriptan + naproxen
  Interventions: Drug: naratriptan + naproxen
- naratriptan (Active Comparator)
  Interventions: Drug: naratriptan
- naproxen (Active Comparator)
  Interventions: Drug: naproxen

INTERVENTIONS:
Drug: naratriptan + naproxen — Tablets containing naratriptan 2,5 mg + naproxen 500 mg
  Arms: naratriptan + naproxen
Drug: naratriptan — Tablets containing naratriptan 2,5 mg
  Arms: naratriptan
Drug: naproxen — Tablets containing naproxen 500 mg
  Arms: naproxen

SUMMARY:
The purpose of this study is to determine whether a fixed-dose combination of naratriptan 2,5 mg + naproxen 500 mg is effective and safe compared each monotherapy for the acute treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, age in the range of 18-65 years inclusive that has onset of migraine before age 50;
* Patient has at least a 3-month history of migraine with or without aura according to the ICHD-II, 2004, IHS (International Headache Society) criteria;
* Patients experienced an average migraine headache frequency of 2-6 moderate or severe attacks per month in the last 03 months prior to screening visit;
* Patients able to distinguish his/her migraine attacks from any other types of headaches;
* Patients able to understand and consent to participate in this clinical study, expressed by signing the Informed Consent (IC).

Exclusion Criteria:

* History of more than 6 migraine attacks/month in the last 03 months prior to screening visit;
* History of non-migraine headache frequency ≥ 15 days/month in each of the 3 months prior to screening;
* History of following migraine variants, according to the ICHD-II, 2004, IHS (International Headache Society): basilar migraine, aura without headache, familial hemiplegic migraine, sporadic hemiplegic migraine or aura with non-migraine headache;
* If female of childbearing potential, has a negative urine pregnancy test at Visit 0 and doesn't use, or doesn't agree to use, for the duration of the study, a medically acceptable form of contraception as determined by the investigator;
* Woman in pregnancy or lactation period;
* History of epilepsy or psychiatric condition that may affect the compliance of the treatment;
* Patients in acupuncture treatment for the symptoms of migraine attacks;
* History or symptoms of cardiovascular disease (myocardial infarction, ischemic heart disease, or with Prinzmetal's angina) or has symptoms of ischemic heart disease;
* Suffers from peripheral vascular disease;
* History of cerebrovascular pathology including stroke and/or transient ischemic attacks;
* History of allergic reactions to naproxen preparations, including subjects in whom aspirin or other NSAID drugs induce the syndrome of asthma, rhinitis, nasal polyps or urticaria;
* Diagnosis of renal or hepatic failure;
* Has significant (as determined by the investigator) cardiovascular risk factors that may include uncontrolled high blood pressure, post-menopausal women, males over 40 years old, hypercholesterolemia, obesity, diabetes mellitus, smoking, or a family history of cardiovascular disease in a 1st degree relative;
* Patients who have stopped or changed the dosage of the preventive treatment of migraine in the last 2 weeks prior the screening visit (V0), including the use of calcium channel blockers, tricyclic antidepressants, beta blockers or serotonergic medications for any other indications;
* Use of prohibited medicine as shown in 9.3 item of this protocol;
* Inability to understand and report the categorical scale debilitating functional of study or symptoms diary;
* Has abused, in the opinion of the Investigator, any of the following drugs, currently or within the past 2 years: opioids, alcohol, barbiturates, benzodiazepine, cocaine or abuse of drugs for migraine treatment including narcotics or ergotamines headache in the past 03 months;
* Hypersensitivity to naratriptan, naproxen, or any of its components;
* Hypersensitivity to sulfonamides;
* History of malignancy ≤ 5 years or > 5 years without documentation of remission / cure, for example, melanoma, leukemia, lymphoma, myeloproliferative disorders and renal cell carcinoma of any duration. Exception: Subjects with basal cell skin cancers, squamous cell, and cervical cancer in situ may be eligible;
* Participation in last one year of clinical protocols, unless it can be direct benefit to patient;
* Any finding of clinical observation (anamnesis and physical exam) laboratory abnormality (eg, blood glucose, blood count), disease (for example, liver, cardiovascular system, lung) or therapy that, in opinion of the investigator, may endanger the patient or interfere with the endpoints of study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Headache relief 2 hours after dosing, without use of rescue medication | 2 hours after single dose treatment
  Participants were evaluated (self-assessment) for pain intensity by using a 4-point rating scale: 0= none, 1= mild, 2= moderate, and 3= severe.

SECONDARY OUTCOMES:
Headache relief 4 hours after dosing, without use of rescue medication | 4 hours after single dose treatment
  Participants were evaluated (self-assessment) for pain intensity by using a 4-point rating scale: 0= none, 1= mild, 2= moderate, and 3= severe
Maintenance of pain relief between 2 and 24 hours after dosing, without use of rescue medication | 2 to 24 hours after single dose treatment
  Participants were evaluated (self-assessment) for pain intensity by using a 4-point rating scale: 0=none, 1=mild, 2=moderate, and 3=severe.
Pain-free response 2 and 4 hours after dosing, without use of rescue medication | 2 and 4 hours after single dose treatment
  Participants were evaluated (self-assessment) for pain intensity by using a 4-point rating scale: 0= none, 1= mild, 2= moderate, and 3= severe.
Maintenance of pain-free response between 2 and 24 hours, without use of rescue medication | 2 to 24 hours after single dose treatment
  Participants were evaluated (self-assessment) for pain intensity by using a 4-point rating scale: 0= none, 1= mild, 2= moderate, and 3= severe.
Freedom from nausea, vomiting, photophobia and phonophobia 2 and 4 hours after dosing | 2 and 4 hours after single dose treatment
  Participants were evaluated (self-assessment) for the presence of vomiting, nausea, photophobia and phonophobia.
Maintenance of freedom from nausea, vomiting, photophobia and phonophobia between 2 and 24 hours after dosing, without use of rescue medication | 2 to 24 hours after single dose treatment
  Participants were evaluated (self-assessment) for the presence of vomiting, nausea, photophobia and phonophobia.
Recurrence of pain between 2 and 24 hours after dosing, without use of rescue medication | 2 to 24 hours after single dose treatment
  Participants were evaluated (self-assessment) for pain intensity by using a 4-point rating scale: 0= none, 1= mild, 2= moderate, and 3= severe.
Proportion of subjects who used rescue medication between 2 and 24 hours after dosing, at least once | 2 to 24 hours after single dose treatment
  Participants were evaluated (self-assessment) about use of rescue medication.
Safety descriptive about occurence of adverse events, evaluation of results of general physical examination. | Collection of safety data throughout the whole study period